CLINICAL TRIAL: NCT06479330
Title: Evaluating the Impact of Incremental Doses of a Sugar Replacer Blend on Gastrointestinal Tolerance in Chocolate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KBE070 / INQ-2402
Record Dates: First submitted 2024-06-19; First posted 2024-06-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Tolerance; Healthy Population
Keywords: sugar replacers; gastrointestinal symptoms; Bowel Habits Diary - Bristol Stool Scale (BHD-BSS); Gastrointestinal Tolerance Questionnaire (GITQ); Acute; Chocolate

STUDY DESIGN:
Intervention Model Description: In a 5-way cross-over, there is a set of 10 balanced sequences to which participants will be randomly assigned. Blocks of 1 or 2 sets of sequences will be randomly ordered to create a balanced sequence for n=60 participants. Orders will be assigned to participants in the order they attended for the first visit after being recruited.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The products will be labelled with a code so study staff and research participants will be blinded as to which test meal is which. After the database will be cleaned and locked, and statistical analysis will be completed, and the codes will be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control chocolate with sugar (Placebo Comparator): Milk chocolate made with sugar at a dose of 45 g (2 servings)
  Interventions: Other: Milk Chocolate
- Maltitol chocolate (Active Comparator): Milk chocolate with maltitol replacing all sugar at a dose of 45 g (2 servings)
  Interventions: Other: Milk Chocolate
- Kestose chocolate (Active Comparator): Milk chocolate with kestose oligofructose replacing all sugar at a dose of 45 g (2 servings)
  Interventions: Other: Milk Chocolate
- Kestose + cocoa and polydextrose premix dose 1 chocolate (Active Comparator): Millk chocolate with kestose oligofructose + cocoa and polydextrose premix dose 1 replacing all sugar at a dose of 45 g (2 servings)
  Interventions: Other: Milk Chocolate
- Kestose + cocoa and polydextrose premix dose 2 chocolate (Active Comparator): Millk chocolate with kestose oligofructose + cocoa and polydextrose premix dose 2 replacing all sugar at a dose of 45 g (2 servings)
  Interventions: Other: Milk Chocolate

INTERVENTIONS:
Other: Milk Chocolate — Acute intake

SUMMARY:
This study is a randomized, double-blind, crossover trial aiming at evaluating the gastrointestinal tolerance of sugar replacer ingredients and blends (maltitol, kestose (Oligofructose), kestose + cocoa and polydextrose premix at different doses)

DETAILED DESCRIPTION:
The study will have a randomized, double-blind, crossover design with 5 visits consisting of one screening visit and 5 study visits (3-14-day interval between the start of each visit) across 2-8 weeks. Participants will be randomized to a test sequence and will consume one control product and 4 test products made with the sugar replacer ingredients or blend of ingredients over the course of the study. At each visit, eligible participants will come to the lab between 8-11am, and ~1-2 hours after consuming their usual breakfast at home. After rating the severity of gastrointestinal symptoms, participants will consume one of the investigational products with a drink of water (250ml) and then be free to leave. The severity of 8 gastrointestinal symptoms (abdominal bloating, abdominal pain, flatulence, burping, reflux (heartburn), stomach rumbling (borborygmus), nausea and vomiting) will be rated at 2, 4, 6, 10 and 24 hours after starting to eat. Over the 24 hour period following consuming the investigational product a Bowel Habit Diary will be kept. For each bowel movement passed during the 24 hour period, participants will be asked to record: the time, if they had to strain, if they experienced discomfort, if they felt there was incomplete evacuation and the consistency of the stool rated using the Bristol Stool Scale (BSS).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, healthy individuals aged 18-55 years, inclusive
* Body Mass Index (BMI) 18.5-32.0kg/m², inclusive
* No major illness, trauma or surgery requiring hospitalization within 3 months of the screening visit
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Non-smokers or smokers who smoke <10 cigarettes/day and are willing not to change nicotine habits during the study period
* Willing to limit alcohol consumption to ≤3 standard drinks/day and ≤7 standard drinks/week during the study period
* Willing to refrain from any marijuana or hemp products during the study period
* Normal bowel habits (>2 bowel movements/week and <3 bowel movements per day)
* Consumes ≤4 servings/day of fruits and vegetables combined and ≤3 (women) or ≤4 (men) servings/day of whole grains using the definitions of "serving" .
* Participants must have a cell phone/tablet/computer and be willing and able to use it to collect study data
* Participants must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP (Ontario Health Insurance Plan)
* Participants are willing to follow current COVID guidelines with respect to attending study visits

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Chronic moderate to severe gastrointestinal symptoms
* Use of systemic antibiotics, antifungals or antiparasitics in the past 3 months and during the experimental period
* Use of medications, supplements, and products which may affect the results (laxative, anti-diarrhea, anti-constipation drugs, high fiber supplements)
* Individuals with any medical conditions or use of supplements or medications that increase risk to the subject or others or may affect the results, as judged by the Principal - Investigator
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Total Area Under the Curve (tAUC) of composite gastrointestinal Symptom score | tAUC between 0 and 24 hours
  total area under the curve (tAUC) of the composite GastroIntestinal symptom score (sum of the scores for the 8 GI symptoms). The score values can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions).

SECONDARY OUTCOMES:
Total Area Under the Curve of each individual gastrointestinal symptom | tAUC between 0 and 24 hours
  Total Area Under the Curve of each of the individual 8 gastrointestinal symptoms (abdominal bloating, abdominal pain, flatulence, burping, reflux, stomach rumbling, nausea, vomiting). Each symptom range from 0 up to 3 with 3 showing the highest / worse condiiton of symptoms
Frequency of composite score > 1 at each time point | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants who have a composite GastoInestinal symptom score >1 (moderate-to-severe) at each time point. The composite score can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions)
Frequency of Diarrhea within 24 hours | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants with diarrhea, defined as 3 or more type 6 or 7 stools (based on the BSS) within the 24 hour period after consumption of the study products
Time for maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time of maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Number of bowel movements | Evaluation performed over 24 hour after consumption of study products
  Number of bowel movements over the 24 hours
straining during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having to strain or not
discomfort during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having discomfort or not
incomplete evacuation | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants declaring incomplete evacuation or not
Stool consistency based on bristol stool scale | Evaluation performed over 24 hour after consumption of study products
  mean stool consistency on Bristol Stool Scale (BSS). The scale provide values from 1 to 7 depending on the type of stool with 1 being the driest stools and 7 the most liquid one.

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No